CLINICAL TRIAL: NCT05056987
Title: Clinical Assessment of Two Daily Wear Reusable Soft Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CLY935-C018
Record Dates: First submitted 2021-09-15; First posted 2021-09-27 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Refractive Errors
Keywords: Contact Lenses; Myopia
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TOTAL30, then AOHP (Other): Lehfilcon A contact lenses worn first, with senofilcon A contact lenses worn second, as randomized. The lehfilcon A contact lenses will be worn for approximately 28 days. The senofilcon A contact lenses will be worn for approximately 14 days. Lenses will be worn bilaterally (in both eyes) in a daily wear modality, with AOSEPT PLUS with HydraGlyde used for nightly cleaning and disinfection.
  Interventions: Device: Lehfilcon A contact lenses; Device: Senofilcon A contact lenses; Device: AOSEPT PLUS with HydraGlyde
- AOHP, then TOTAL30 (Other): Senofilcon A contact lenses worn first, with lehfilcon A contact lenses worn second, as randomized. The senofilcon A contact lenses will be worn for approximately 14 days. The lehfilcon A contact lenses will be worn for approximately 28 days. Lenses will be worn bilaterally (in both eyes) in a daily wear modality, with AOSEPT PLUS with HydraGlyde used for nightly cleaning and disinfection.
  Interventions: Device: Lehfilcon A contact lenses; Device: Senofilcon A contact lenses; Device: AOSEPT PLUS with HydraGlyde

INTERVENTIONS:
Device: Lehfilcon A contact lenses — CE-marked spherical soft contact lenses worn according to to the product package insert/Instructions for Use
  Other Names: TOTAL30®
Device: Senofilcon A contact lenses — CE-marked spherical soft contact lenses worn according to to the product package insert/Instructions for Use
  Other Names: ACUVUE OASYS® with HYDRACLEAR® Plus; AOHP
Device: AOSEPT PLUS with HydraGlyde — Hydrogen peroxide-based cleaning and disinfecting solution
  Other Names: AOSEPT® PLUS with HYDRAGLYDE®

SUMMARY:
The overall objective of this clinical study is to describe the clinical performance of the TOTAL30® soft contact lens compared to the ACUVUE® OASYS® with HYDRACLEAR PLUS (AOHP) soft contact lens in a daily wear modality.

DETAILED DESCRIPTION:
Subjects will be expected to attend 3 visits and wear the study contact lenses at least 5 days per week and at least 8 hours per day. On Visits 2 and 3, subjects will be expected to wear the study lenses at least 6 hours prior to the study visit. The expected total duration of subject participation in the study will be approximately 1.5 months. This study will be conducted in the United Kingdom (UK).

ELIGIBILITY:
Key Inclusion Criteria:

* Currently wearing any commercial spherical soft contact lenses with at least 3 months wearing experience.
* Willing to wear the study lenses for a minimum of 5 days per week and 8 hours per day.
* Willing to NOT use rewetting/lubricating drops at any time during the study.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Participation in a clinical trial within the previous 14 days or currently enrolled in any clinical trial.
* Habitual AOHP contact lens wearers (in the past 3 months).
* Monovision wear during the study.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (1):
- Eurolens Research, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one investigative site located in the United Kingdom.
Pre-assignment Details: This reporting group includes all enrolled subjects/eyes.
Units Other Than Participants: eyes
Groups:
- TOTAL30, Then AOHP: Lehfilcon A contact lenses worn first, with senofilcon A contact lenses worn second, as randomized. The lehfilcon A contact lenses were worn for approximately 28 days. The senofilcon A contact lenses were worn for approximately 14 days. Lenses were worn bilaterally (in both eyes) in a daily wear modality, with AOSEPT PLUS with HydraGlyde used for nightly cleaning and disinfection.
- AOHP, Then TOTAL30: Senofilcon A contact lenses worn first, with lehfilcon A contact lenses worn second, as randomized. The senofilcon A contact lenses were worn for approximately 14 days. The lehfilcon A contact lenses were worn for approximately 28 days. Lenses were worn bilaterally (in both eyes) in a daily wear modality, with AOSEPT PLUS with HydraGlyde used for nightly cleaning and disinfection.
Period: First Wear Period, Day 14 or Day 28
Arm/Group | TOTAL30, Then AOHP | AOHP, Then TOTAL30
Started | 18; 36 eyes | 18; 36 eyes
Completed | 17; 34 eyes | 16; 32 eyes
Not Completed | 1; 2 eyes | 2; 4 eyes
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Period: Second Wear Period, Day 14 or Day 28
Arm/Group | TOTAL30, Then AOHP | AOHP, Then TOTAL30
Started | 17; 34 eyes | 16; 32 eyes
Completed | 17; 34 eyes | 16; 32 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | TOTAL30, Then AOHP | AOHP, Then TOTAL30 | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (11.3) | 32.9 (10.6) | 30.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 7 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Distance VA (logMAR) With Study Lenses
Description: Distance visual acuity (VA) was assessed for each eye individually with study lenses in place using letter charts. VA was measured in logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with lower logMAR values indicating better visual acuity. The follow-up visit for TOTAL 30 occurred approximately 28 days after the baseline visit. The follow-up visit for AOHP occurred approximately 14 days after the baseline visit. No formal hypothesis was formulated for the primary effectiveness endpoint of distance VA; hence, no inferential testing was performed.
Time Frame: Dispense (Day 0) and Follow-Up (Day 28 for TOTAL30, Day 14 for AOHP) (each wear period)
Population: Safety analysis set: All subjects/eyes exposed to any study lenses evaluated in this study with non-missing responses.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- TOTAL30: Lehfilcon A contact lenses worn in Period One or Period 2, as randomized. The lenses were worn for approximately 28 days bilaterally (in both eyes) in a daily wear modality, with AOSEPT PLUS with HydraGlyde used for nightly cleaning and disinfection.
- AOHP: Senofilcon A contact lenses worn in Period One or Period 2, as randomized. The lenses were worn for approximately 14 days bilaterally (in both eyes) in a daily wear modality, with AOSEPT PLUS with HydraGlyde used for nightly cleaning and disinfection.
Arm/Group | TOTAL30 | AOHP
Number analyzed (Participants) | 34 | 35
Number analyzed (eyes) | 68 | 70
logMAR
  Dispense | -0.08 (0.07) | -0.10 (0.07)
  Follow Up: number analyzed (Participants) | 33 | 34
  Follow Up: number analyzed (eyes) | 66 | 68
  Follow Up | -0.07 (0.09) | -0.07 (0.07)

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 1.5 months.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of participants. This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Pretreatment: Events reported in this group occurred prior to dispense of the study contact lenses
- TOTAL30 Ocular; TOTAL30 Non-ocular: Events reported in this group occurred following dispense of the lehfilcon A contact lenses
- AOHP Ocular; AOHP Non-ocular: Events reported in this group occurred following dispense of the senofilcon A contact lenses
Arm/Group | Pretreatment | TOTAL30 Ocular | TOTAL30 Non-ocular | AOHP Ocular | AOHP Non-ocular
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/68 | 0/34 | 0/70 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/68 | 0/34 | 0/70 | 0/35
Other Adverse Events (participants affected / at risk) | 0/36 | 0/68 | 0/34 | 0/70 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT05056987/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT05056987/SAP_001.pdf